CLINICAL TRIAL: NCT06207344
Title: The Anesthesia Effects of Dexmedetomidine Combined With Desflurane or Propofol in Lobectomy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Bing Chen, Ph.D, Associate professor, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023.159
Record Dates: First submitted 2023-10-26; First posted 2024-01-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Anesthesia Recovery Period; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Dexmedetomidine; Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine and propofol (Active Comparator): After anesthesia induction, dexmedetomidine was infused intravenously at 1 μg/kg within 15 min, then infused at 0.3 μg/kg/h until 30 min before the end of the operation. Propofol was infused intravenously at 4-12mg/kg/h to maintain the depth of anesthesia (patient state index between 25-50 monitored by Masimo SedLine).
  Interventions: Drug: Dexmedetomidine and propofol
- Dexmedetomidine and desflurane (Experimental): After anesthesia induction, dexmedetomidine was infused intravenously at 1 μg/kg within 15 min, and then infused at 0.3 μg/kg/h until 30 min before the end of the operation. At the same time, 2.5%-8.5% desflurane was used to maintain the depth of anesthesia (patient state index between 25-50 monitored by Masimo SedLine).
  Interventions: Drug: Dexmedetomidine and desflurane

INTERVENTIONS:
Drug: Dexmedetomidine and propofol — Group 1: After anesthesia induction, dexmedetomidine was infused at 1 μg/kg intravenously within 15 min, then infused at 0.3 μg/kg/h until 30 min before the end of the operation. Meantime, propofol was infused at 4-12mg/kg/h intravenously to maintain the depth of anesthesia.
  Other Names: Dexmedetomidine Hydrochloride injection and propofol injectable emulsion
  Arms: Dexmedetomidine and propofol
Drug: Dexmedetomidine and desflurane — Group 2: After anesthesia induction, dexmedetomidine was infused at 1 μg/kg intravenously within 15 min, then infused at 0.3 μg/kg/h until 30 min before the end of the operation. At the same time, 2.5%-8.5% desflurane was inhaled to maintain the depth of anesthesia.
  Other Names: Dexmedetomidine Hydrochloride injection and Suprane
  Arms: Dexmedetomidine and desflurane

SUMMARY:
In one-lung ventilation surgery, compared with dexmedetomidine combined with propofol, dexmedetomidine combined with desflurane may be beneficial to accelerate patients' recovery and reduce postoperative pulmonary complications and does not increase the incidences of delirium and postoperative nausea and vomiting.

DETAILED DESCRIPTION:
With the increase in the prevalence of lung cancer in recent years, the number of patients undergoing lobectomy has also increased. When performing lobectomy, inserting a double-lumen endotracheal tube or bronchial occlusive device and then ventilating the healthy lung is necessary. The affected lung is not ventilated; that is one-lung ventilation, which can fully expose the vision of the affected lung, provide space for surgical operation, and simultaneously avoid the pollution of the healthy lung. The emergence of one-lung ventilation has extensively promoted the development of thoracic surgery. However, during one-lung ventilation, the affected lung is not ventilated, and the blood flow of the affected lung is not oxygenated, which leads to increased intrapulmonary shunt and hypoxemia. Repeated and excessive inflation of the healthy lung may release many inflammatory factors, trigger local or systemic inflammatory reactions, and increase postoperative pulmonary complications. Therefore, it is an essential goal of anesthesia management to quickly wake up and resume spontaneous breathing to reduce mechanical ventilation time.

Propofol-based intravenous anesthesia and inhalation anesthesia with sevoflurane, isoflurane, or desflurane are clinics' most commonly used general anesthesia methods. It is found that inhalation anesthesia with desflurane is superior to propofol-based intravenous anesthesia in the aspects of eye-opening time, spontaneous breathing recovery time, and extubation time in outpatient surgery, lung volume reduction surgery, lung cancer surgery, and endoscopic lumbar disc surgery. In addition, several meta-analyses found that inhalation anesthesia has an anti-inflammatory effect compared with propofol-based anesthesia, which can reduce alveolar inflammatory reaction and postoperative pulmonary complications in patients with one-lung ventilation. Kawanishi et al. found that desflurane inhalation anesthesia can promote the collapse of the affected lung, shorten the operation time, and reduce the occurrence of atelectasis compared with propofol-based intravenous anesthesia. These studies show that inhalation anesthesia with desflurane is superior to propofol-based intravenous anesthesia in one-lung ventilation surgery.

However, inhalation anesthesia is not perfect, and studies have also found that inhalation anesthesia increases the incidences of restlessness during awakening and postoperative nausea and vomiting. One study found that the incidences of delirium, nausea and vomiting in the desflurane anesthesia group were 50% and 37.5% respectively, while that in the propofol-based intravenous anesthesia group was 10% and 17.5% respectively in lung cancer surgery. Therefore, it is necessary to explore an anesthesia management method that will not affect the advantages of inhalation anesthesia but also reduce the disadvantages of inhalation anesthesia.

Dexmedetomidine is a highly selective α2- adrenergic receptor agonist. Its primary function is sedation, often used as an anesthetic adjuvant. Studies have found that dexmedetomidine can significantly reduce the incidences of delirium during recovery and postoperative nausea and vomiting. In patients undergoing nasal surgery, dexmedetomidine can reduce the incidence of delirium in patients receiving desflurane anesthesia from 52.8% to 5.6%, even lower than the incidence of delirium (10%) in patients receiving propofol in lung cancer surgery. In patients undergoing laparoscopic hysterectomy, the use of dexmedetomidine can reduce the incidence of nausea and vomiting after desflurane anesthesia from 32% to 13%, even lower than that after propofol anesthesia in lung cancer surgery (17.5%). In addition, dexmedetomidine can reduce inflammatory reactions, improve oxidative stress and respiratory mechanics, reduce intrapulmonary shunt, improve oxygenation, and reduce postoperative pulmonary complications in one-lung ventilation surgery. Although dexmedetomidine has a sedative effect, this sedative effect can be awakened easily. Moreover, a meta-analysis found that dexmedetomidine did not prolong the stay time in the anesthesia recovery room but only prolonged extubation time statistically, and it had no clinical significance. In a word, a large number of meta-analyses found that dexmedetomidine can not only reduce the incidence of various adverse events after operation but also has no noticeable effect on patients' recovery.

Therefore, the investigators speculate that compared with dexmedetomidine combined with propofol, dexmedetomidine combined with desflurane is beneficial to accelerate patients' recovery and reduce postoperative pulmonary complications and does not increase the incidences of delirium and postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective thoracoscopic unilateral lobectomy.
2. General anesthesia is required and the expected duration of one-lung ventilation is ≥ 1h.
3. American Association of Anesthesiologists (ASA) physical condition classification I-III.
4. Patients over 18 years old.
5. Voluntary participation and ability to understand and sign the informed consent.

Exclusion Criteria:

1. Obese patients (BMI>28 kg/m2).
2. patients with grade 3 hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg).
3. Acute coronary syndrome, sinus bradycardia (heart rate < 45 beats/min), II or III degree atrioventricular block, NYHA heart function classification III or IV.
4. Patients with severe history of chronic obstructive pulmonary disease (GOLD grade III or IV of pulmonary function of chronic obstructive pulmonary disease), severe or uncontrolled bronchial asthma, pulmonary infection, bronchiectasis and thoracic deformity.
5. Pulmonary artery pressure ≥60 mmHg.
6. Patients with Child grade B or C of liver function.
7. Patients with chronic kidney disease in stage 4 or 5.
8. Patients with hyperthyroidism and pheochromocytoma.
9. Patients who are expected to need mechanical ventilation after operation.
10. People with hearing, intelligence, communication and cognitive impairment.
11. For any reason, it is impossible to cooperate with the study or the researcher thinks that it is not suitable to be included in this experiment.
12. patients who are expected to be transferred to ICU after operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-21 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to open eyes after anesthetics withdrawal | From time of anesthetic withdrawal to the first time of the patient open his or her eyes, assessed up to 2 hour.
  The first time to open eyes after anesthetics withdrawal.

SECONDARY OUTCOMES:
Incidence of delirium | From time of anesthetic withdrawal to the patient leaving the postanesthesia care unit, assessed up to 2 hour.
  The Richmond Agitation-Sedation Scale (RASS) will be used to assess the incidence of delirium. RASS is a 10-point scale, with four levels of anxiety or agitation (+1 to +4 [combative]), one level to denote a calm and alert state (0), and 5 levels of sedation (-1 to -5) culminating in unarousable (-5). The scores of +2, +3, and +4 are defined as delirium.
Incidence of nausea and vomiting | From time of anesthetic withdrawal to the patient leaving the postanesthesia care unit, assessed up to 2 hour.
  The severity of nausea and vomiting will be evaluated by visual analogue scale (VAS): a 10 cm ruler was used as a scale, one end (0 points) indicated no nausea and vomiting, and the other end was 10 cm, indicating the most severe nausea and vomiting that was unbearable (1~4 was mild, 5~6 was moderate, and 7~10 was severe).
Pain level | From time of anesthetic withdrawal to the patient leaving the postanesthesia care unit, assessed up to 2 hour.
  Numeric Rating Scale will be used to assess the degree of pain. 0~10 is used to represent different degrees of pain: 0 is no pain, 1~3 is mild pain (the pain does not affect sleep), 4~6 is moderate pain (mildly affects sleep), 7~9 is severe pain (unable to fall asleep or wakes up from sleep), and 10 is severe pain.
Incidences of other side effects | From time of anesthetic withdrawal to the patient leaving the postanesthesia care unit, assessed up to 2 hour.
  Any unquestioned side effects will be recorded, such non-planned intensive care unit transfer, unplanned reoperation, unplanned reintubation, etc.
Drugs and their dosage | From time of anesthetic withdrawal to the patient leaving the postanesthesia care unit, assessed up to 2 hour.
  These drugs and their dosage will be recorded, such as muscle relaxant antagonism, antiemetic drugs, and analgesic drugs.
QoR-40 scores | Postoperative day 1 and 3.
  QoR-40 scores will be used to assess the quality of recovery. The questionnaire consists of five subscales: emotional status (9 items), physical comfort (12 items), psychological support (7 items), physical independence (5 items), and pain (7 items). All the items are rated on a five-point scale ranging from 1 to 5. The initial point and conversion score of each item are calculated. Depending on the question, the best answers may have a score of either 5 or 1. The best answers to positive questions are scored 5, while the best answers to negative questions are assigned the score of 1. The total score of QoR-40 is given by the summation of scores for all items and ranges from 40 to 200. The higher the score, the better is the health status.Citation
Postoperative pulmonary complications | First 7 postoperative days
  The incidence of postoperative pulmonary complications was assessed according to the Assess Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) definition. The severity of postoperative pulmonary complications was scored on a 0-5 scale.
White blood cell count | Postoperative day 1 and 3.
  White blood cell count will be used to assess the inflammatory level.
Neutrophil ratio | Postoperative day 1 and 3.
  Neutrophil ratio will be used to assess the inflammatory level.
Lymphocyte ratio | Postoperative day 1 and 3.
  Lymphocyte ratio will be used to assess the inflammatory level.
C-reactive protein | Postoperative day 1 and 3.
  C-reactive protein will be used to assess the inflammatory level.
Time for tidal volume of spontaneous breathing over 300 ml | From time of anesthetic withdrawal to the patient tidal volume of spontaneous breathing over 300 ml, assessed up to 2 hour.
  Time from anesthetics withdrawal to tidal volume of spontaneous breathing over 300 ml.
Extubation time | From time of anesthetic withdrawal to the tracheal tube was extubated, assessed up to 2 hour.
  Time from anesthetics withdrawal to extubation
Postanesthesia care unit residence time | From time of anesthetic withdrawal to the patient leaving the postanesthesia care unit, assessed up to 2 hour.
  Time of staying in postanesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Bing Chen, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available with the responding author when required.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available when publish and keep it for 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Campos JH, Feider A. Hypoxia During One-Lung Ventilation-A Review and Update. J Cardiothorac Vasc Anesth. 2018 Oct;32(5):2330-2338. doi: 10.1053/j.jvca.2017.12.026. Epub 2017 Dec 19. No abstract available. PMID 29361458
- [Background] Bernasconi F, Piccioni F. One-lung ventilation for thoracic surgery: current perspectives. Tumori. 2017 Nov 23;103(6):495-503. doi: 10.5301/tj.5000638. Epub 2017 Jun 7. PMID 28604996
- [Background] Karzai W, Haberstroh J, Priebe HJ. Effects of desflurane and propofol on arterial oxygenation during one-lung ventilation in the pig. Acta Anaesthesiol Scand. 1998 Jul;42(6):648-52. doi: 10.1111/j.1399-6576.1998.tb05296.x. PMID 9689269
- [Background] Abe K, Shimizu T, Takashina M, Shiozaki H, Yoshiya I. The effects of propofol, isoflurane, and sevoflurane on oxygenation and shunt fraction during one-lung ventilation. Anesth Analg. 1998 Nov;87(5):1164-9. doi: 10.1097/00000539-199811000-00035. PMID 9806702
- [Background] Cho YJ, Kim TK, Hong DM, Seo JH, Bahk JH, Jeon Y. Effect of desflurane-remifentanil vs. Propofol-remifentanil anesthesia on arterial oxygenation during one-lung ventilation for thoracoscopic surgery: a prospective randomized trial. BMC Anesthesiol. 2017 Jan 18;17(1):9. doi: 10.1186/s12871-017-0302-x. PMID 28100177
- [Background] Kawanishi R, Kakuta N, Sakai Y, Hari Y, Sasaki H, Sekiguchi R, Tanaka K. Desflurane improves lung collapse more than propofol during one-lung ventilation and reduces operation time in lobectomy by video-assisted thoracic surgery: a randomized controlled trial. BMC Anesthesiol. 2022 Apr 29;22(1):125. doi: 10.1186/s12871-022-01669-7. PMID 35488195
- [Background] Yuan JL, Kang K, Li B, Lu J, Miao MR, Kang X, Zhang JQ, Zhang W. The Effects of Sevoflurane vs. Propofol for Inflammatory Responses in Patients Undergoing Lung Resection: A Meta-Analysis of Randomized Controlled Trials. Front Surg. 2021 Jul 2;8:692734. doi: 10.3389/fsurg.2021.692734. eCollection 2021. PMID 34277696
- [Background] Jannu V, Dhorigol MG. Effect of Intraoperative Dexmedetomidine on Postoperative Pain and Pulmonary Function Following Video-assisted Thoracoscopic Surgery. Anesth Essays Res. 2020 Jan-Mar;14(1):68-71. doi: 10.4103/aer.AER_9_20. Epub 2020 Mar 16. PMID 32843795
- [Background] Jiang H, Kang Y, Ge C, Zhang Z, Xie Y. One-lung ventilation patients: Clinical context of administration of different doses of dexmedetomidine. J Med Biochem. 2022 Apr 8;41(2):230-237. doi: 10.5937/jomb0-33870. PMID 35510198
- [Background] Xia R, Xu J, Yin H, Wu H, Xia Z, Zhou D, Xia ZY, Zhang L, Li H, Xiao X. Intravenous Infusion of Dexmedetomidine Combined Isoflurane Inhalation Reduces Oxidative Stress and Potentiates Hypoxia Pulmonary Vasoconstriction during One-Lung Ventilation in Patients. Mediators Inflamm. 2015;2015:238041. doi: 10.1155/2015/238041. Epub 2015 Jul 26. PMID 26273134